CLINICAL TRIAL: NCT06330636
Title: The Acute Effect of D-allulose Consumption on Postprandial Glycaemia in Healthy Individuals
Brief Title: The Acute Effect of D-allulose Consumption on Postprandial Glycaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Principal Investigator, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 336-0723
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Sugar; Blood, High
Keywords: glycaemia response; D-allulose; dietary carbohydrates
MeSH Terms: conditions — Hyperglycemia | interventions — Saccharin

STUDY DESIGN:
Intervention Model Description: Randomised, placebo controlled cross over design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Allocation coded A and B, with independent researcher determining allocation and making up the test breakfasts for the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-Allulose (Experimental): 15g D-Allulose added to a high glycaemic index oat porridge
  Interventions: Other: D-Allulose
- Saccharin (Placebo Comparator): Sodium saccharin (1x 'Sweetex' tablet) added to a high glycaemic index oat porridge
  Interventions: Other: Sodium Saccharin

INTERVENTIONS:
Other: D-Allulose — Test breakfast
  Other Names: Test Day
  Arms: D-Allulose
Other: Sodium Saccharin — placebo breakfast
  Other Names: Control Day
  Arms: Saccharin

SUMMARY:
The rare sugar D-Allulose, when consumed in a drink before eating has been shown to reduce the blood glucose response to high carbohydrate drinks or meals in people who are healthy, or have elevated fasting blood glucose concentration. However, the effectiveness of D-allulose to suppress blood glucose concentration when added into carbohydrate containing food products has not been previously reported and as the potential use of allulose is as a sucrose replacer in foods, rather than drinks, it is important that effects and efficacy are tested in this format. The study aimed to extend understanding of the acute effects of D-allulose consumption in humans by testing whether post-eating blood glucose concentration can be modified by the presence of D-allulose in a high carbohydrate breakfast and collecting data on any adverse gastrointestinal effects of consuming D-allulose.

DETAILED DESCRIPTION:
Twelve healthy individuals (age 18-40y, BMI 19-30 kg/m2) will be recruited following a health screening. An equal number of males and females will be sought to improve generalisability of data, but the study will not powered to explore sex differences in response. After a successful screening and recruitment, participants will be asked to record everything that they eat and drink in a dietary record for 4 days (3 week and 1 weekend day). This will be analysed using dietary analysis software (Nutritics, Eire) for energy, macronutrient and fibre intake to characterise the participants' habitual diets.

At 2 subsequent laboratory visits, volunteers will be asked to refrain from drinking alcohol and doing strenuous exercise on the day before. They will arrive at the laboratory by 9am after an overnight fast and a retrograde cannula will be inserted into a superficial dorsal hand vein after prior intradermal infiltration with ~0.01ml 1% lidocaine. The cannulated hand will be placed into a hot air hand warmer for the duration of the study to allow sampling of arterialised venous blood for assessment of blood glucose and insulin concentration. A 1ml fasting blood sample will be taken and participants will be asked to complete a short questionnaire containing 6 visual analogue scales. Four of these will assess subjective appetite (How full do you feel? How much food do you think that you could eat? How hungry do you feel? How strong is your desire to eat?) with 2 addressing possible gastrointestinal symptoms (How much abdominal pain are you currently feeling? How much intestinal gurgling are you experiencing?). Participants will be asked to evaluate how strong their feelings are by placing a vertical mark along a 100mm horizontal line; 0 representing not experiencing the criterion at that time, and 100 indicating experiencing the greatest degree of that feeling that they could imagine. The combined appetite score (CAS) will be calculated according to standard methods and expressed as incremental change from the score reported at the end of the meal (iCAS).

Once baseline measures have been made, participants will be given a porridge breakfast (50g Ready Brek™, 15g skimmed milk powder, 10g glucose, 200ml hot water) to which has been added 15g of D-allulose or 1 saccharin tablets (Sweetex™). Fifteen grams of D-allulose and 1 Sweetex™ will be approximately equivalent to the sweetness provided by 10g (2 tsp) of sucrose (table sugar). The base porridge will provide 1.1MJ (265 kcal), 47g carbohydrate (29.1g starch, 17.8g sugars), 10.9g protein and 3.7g fat. The saccharin tablets will add no further energy to the breakfast, but the D-allulose will add a further 25kJ (6 kcal) to the porridge. Both porridge meals have the same volume, taste and consistency. Further 1ml blood samples will be taken at 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes after finishing eating breakfast, with the questionnaire completed immediately after eating and at the 20, 40, 60, 90, 120, 150 and 180 minute time points. At 180 minutes, the cannula will be removed, and participants will be offered refreshments before leaving the laboratory. Therefore, the time in the laboratory on each study visit will be ~4 hours and the amount of blood collected will be <20ml.

The second study visit will be scheduled for at least a week after visit 1, and in the time between visits participants will resume their usual diet and lifestyle. At the second visit, the protocol described above will be repeated, but participants will receive the breakfast that they did not receive at visit 1 i.e. if they received the porridge with D-allulose at visit 1, then they will receive the porridge with saccharin at visit 2 and vice versa.

The order in which the breakfasts are given will be randomly allocated according to a predetermined randomisation plan. The randomisation sequence will be generated for males and females separately to ensure a balanced allocation within sex. Individuals will be randomised at the first laboratory visit, with their randomisation number allocated sequentially. Any participants who withdraw from the study will be replaced if time allows.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Not currently taking any medications (using contraceptive medication is acceptable)
* Aged between 18 and 40 years
* Healthy weight or overweight (Body Mass Index 19-30 kg/m2)

Exclusion Criteria:

* Reporting functional gastrointestinal problems, such as irritable bowel syndrome, gastroparesis or reflux
* History of inflammatory bowel diseases such as Crohn's disease or Ulcerative colitis
* Diabetes mellitus
* Surgical resection of gastrointestinal tract.
* Food allergies, intolerances or acceptability issues related to the standard meal, including veganism, lactose intolerance and coeliac disease.
* Following a restricted habitual diet e.g. low carbohydrate, high protein or meal replacement diet
* Following a restrictive dietary pattern e.g. intermittent fasting
* Currently following a reduced-energy diet to control body weight
* Pregnant or breast feeding
* History or current psychiatric illness
* History or current neurological condition (e.g. epilepsy)
* Taking regular medication, including over the counter and prescription drugs; Oral contraception medication and intermittent use of over the counter pain relief is acceptable.
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Incremental area under the curve (iAUC) 180 Glucose Test | 180 minutes after breakfast ingestion
  Incremental area under the curve (180min) for blood glucose on test day
iAUC 180 Glucose Placebo | 180 minutes after breakfast ingestion
  Incremental area under the curve (180min) for blood glucose on placebo day

SECONDARY OUTCOMES:
Glycaemia Test | 180 minutes after breakfast ingestion
  Postprandial glycaemic response to test breakfast
Glycaemia Placebo | 180 minutes after breakfast ingestion
  Postprandial glycaemic response to placebo breakfast
Insulinemia Test | 180 minutes after breakfast ingestion
  Postprandial circulating insulin response to test breakfast
Insulinemia Placebo | 180 minutes after breakfast ingestion
  Postprandial circulating insulin response to placebo breakfast
iAUC 180 Insulin Test | 180 minutes after breakfast ingestion
  Incremental area under the curve (180min) for circulating insulin on test day
iAUC 180 Insulin Placebo | 180 minutes after breakfast ingestion
  Incremental area under the curve (180min) for circulating insulin on placebo day
iCAS Test | 180 minutes after breakfast ingestion
  incremental 'combined appetite score' response following test breakfast (min 0 - max 100) with a higher number indicating greater appetite
iCAS Placebo | 180 minutes after breakfast ingestion
  incremental 'combined appetite score' response following placebo breakfast (min 0 - max 100) with a higher number indicating greater appetite
abdominal discomfort test | 180 minutes after breakfast ingestion
  abdominal discomfort visual analogue score (min 0- max 100 scale) after test breakfast. Greater score indicates greater discomfort
abdominal discomfort placebo | 180 minutes after breakfast ingestion
  abdominal discomfort visual analogue score (min 0- max 100 scale) after placebo breakfast. Greater score indicates greater discomfort
Dietary Fibre | 4 days
  Dietary fibre intake calculated from 4-day dietary records using nutritional database
Carbohydrate % | 4 days
  Dietary carbohydrate intake expressed as a percentage of total energy intake.
Fat % | 4 days
  Dietary fat intake expressed as a percentage of total energy intake.
Protein % | 4 days
  Dietary protein intake expressed as a percentage of total energy intake.
Sugars % | 4 days
  Dietary sugars intake expressed as a percentage of total energy intake.

CONTACTS AND LOCATIONS:
Overall Officials: Liz Simpson, PhD, Principal Investigator — University of Nottingham
Locations (1):
- David Greenfield Human Physiology Laboratories, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised research data will be made available on request to the study PI
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Once published in the public domain. Availability will be for a period of 7 years from publication, after which time all data will be destroyed
Access Criteria: Access will be subject to ethical constraints, the preservation of intellectual property (IP), and written acknowledgement that it is a research collaboration, with data ownership residing with the original research teams.